CLINICAL TRIAL: NCT06231030
Title: Adaptation, Validity and Reliability of "Unidimensional Self-Efficacy Scale for Multiple Sclerosis (USE-MS)" in Turkish
Brief Title: Unidimensional Self-Efficacy Scale for Multiple Sclerosis (USE-MS) Turkish Adaptation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Gazi University (Other); Hacettepe University (Other)
Responsible Party: Principal Investigator, Asli Celik, Lecturer, PT. MSc., Nigde Omer Halisdemir University
Other Study IDs: Gazi University-05.09.2023
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis; Self Efficacy
Keywords: Multiple sclerosis; Self Efficacy; Adaptation; Validity; Reliability
MeSH Terms: conditions — Multiple Sclerosis | interventions — Acclimatization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis Group: Method Description Study data will be collected multicenter. It will be obtained from individuals diagnosed with MS who applied to Niğde Ömer Halisdemir University Training and Research Hospital Neurology Polyclinic and Hacettepe University, Faculty of Medicine, Department of Neurology and referred to Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation.
  Interventions: Other: Validity, Reliability and Adaptation

INTERVENTIONS:
Other: Validity, Reliability and Adaptation — Expanded Disability Status Scale (EDSS) will be applied by a neurologist to determine the disability level of the individuals included in the study. In addition to the USE-MS scale, the GSE questionnaire, MuSiQoL and NFI-MS will be administered by an expert physiotherapist. The questionnaires and scales to be used in the study will be administered by face-to-face interview method twice in total with two weeks intervals. In addition to the USE-MS scale, the GSE questionnaire, MuSiQoL and NFI-MS will be applied. The questionnaires and scales to be used in the study will be administered by face-to-face interview method 2 times in total with a 2-week interval.

SUMMARY:
Multiple Sclerosis (MS) is a chronic, inflammatory, demyelinating, autoimmune disease of the central nervous system. Despite functional limitations and unpredictable disease course, individuals with MS are aimed to maintain different levels of independence according to the level of disability. It is aimed to develop interventions that aim to increase self-efficacy levels and participation in daily life in individuals with this diagnosis. The "Unidimensional Self-Efficacy Scale for Multiple Sclerosis (USE-MS)" is a self-efficacy scale developed specifically for individuals with MS and answered based on patient declaration. The aim of this study is to adapt the "USE-MS" scale into Turkish and to establish its validity and reliability.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic, inflammatory, demyelinating, autoimmune disease of the central nervous system. Despite functional limitations and unpredictable disease course, individuals with MS are aimed to maintain different levels of independence according to the level of disability. It is aimed to develop interventions that aim to increase self-efficacy levels and participation in daily life in individuals with this diagnosis. The "Unidimensional Self-Efficacy Scale for Multiple Sclerosis (USE-MS)" is a self-efficacy scale developed specifically for individuals with MS and answered based on patient declaration. The scale, which consists of 12 questions in total, includes the assessment of the extent to which patients consider themselves competent during the performance of various tasks or activities. The aim of this study is to adapt the "USE-MS" scale into Turkish and to establish its validity and reliability. The study data will be collected multicenter and will be obtained from individuals diagnosed with MS who applied to Niğde Ömer Halisdemir University Training and Research Hospital Neurology Outpatient Clinic and Hacettepe University, Faculty of Medicine, Department of Neurology and referred to Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. Necessary permissions were obtained from all institutions and the scale developers. After the purpose and method of the study were explained to the participants in detail, individuals who voluntarily agreed to participate in the study will be included. The questionnaires and scales to be used in the study will be administered by face-to-face interview method 2 times in total with 2 weeks intervals. Patients' self-efficacy will be assessed with the USE-MS scale and General Self Efficacy (GSE) questionnaires, their quality of life will be assessed with the Multiple Sclerosis International Quality of Life Questionnaire (Multiple Sclerosis Quality of Life-MuSiQoL) and their fatigue will be assessed with the Neurological Fatique Inventory Multiple Sclerosis (NFI-MS). The serial approach method will be used to translate the original NFI-MS questionnaire into Turkish. In order to determine the comprehensibility of the translated text, the Turkish version of the NFI-MS will be administered to 20 individuals with MS and the parts that are not understood will be revised. Since at least 5-10 times the number of items in the questionnaire should be included for factor analysis, the final version of the questionnaire will be applied to individuals diagnosed with MS with at least 60-120 participants. Cronbach's Alpha Reliability coefficient will be used to determine the internal consistency of the questionnaire and Rasch analysis will be applied for internal construct validity analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS by a neurologist,
* Understands and speaks Turkish,
* Individuals who score 18 points or above on the mini-mental status assessment (MMSA) will be included.

Exclusion Criteria:

* Dementia, hearing and/or vision loss,
* Illiterate patients will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients who applied to Nigde Omer Halisdemir University Training and Research Hospital Neurology Clinic or Hacettepe University Faculty of Medicine Neurology Department or who are referred to Gazi University Department of Physiotherapy and Rehabilitation will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
Unidimensional Self-Efficacy Scale for Multiple Sclerosis (USE-MS) | Baseline
  It is a patient-reported self-efficacy assessment scale specific for MS patients. The original scale has been shown to be reliable and valid for self-efficacy assessment in individuals with MS. Total scoring is obtained by summing all 12 items, but items 5, 7-9 and 11 are reverse scored. USE-MS 0: Strongly disagree, 1: Disagree, 2: Undecided, 3: Agree, 4: Strongly agree on a 5-point Likert scale. The higher the score, the better the self-efficacy beliefs of individuals .
General Self-Efficacy Scale | Baseline
  General Self-Efficacy Scale (GSE) has been 20 items. In 1981, it was revised and the number of items was reduced to 10. The questions in the scale are scored according to the answer given as 1: Not at all suitable for me, 2: Somewhat suitable for me, 3: Mostly suitable for me and 4: Completely suitable for me. The total score of the scale varies between 10-40 points. The higher the score, the better the self-efficacy beliefs of individuals.
Multiple Sclerosis Quality of Life-MuSiQoL | Baseline
  The original version consists of 74 questions and there is also a short form consisting of 31 questions. MuSiQoL consists of a total of 9 subgroups including activities of daily living, psychological status, findings, friendships, family relationships, emotional and sexual life, acceptance, coping with the disease and satisfaction with health services. During the assessments, individuals are asked to answer by taking into account their situation in the last 4 weeks. They are asked to mark the option that best expresses themselves from the options of never (0: Never), rarely (1: Occasionally), sometimes (2: Some), frequently (3: Very) and always (4: Very much).
Neurologic Fatigue Inventory-Multiple Sclerosis (NYI-MS) | Baseline
  It is a 23-item questionnaire. It has four sub-dimensions. These are physical (8 items), cognitive (4 items), recovery with diurnal sleep or rest (6 items) and abnormal nocturnal sleep and sleepiness (5 items). The questions in the questionnaire are scored as 0= Strongly disagree, 1= Disagree, 2= Agree, 3= Strongly agree. Each of the four subscales is calculated separately. However, a total scoring is not made by adding them all together. A high score indicates that the fatigue of the patients is high.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline
  MMSE will be used to evaluate cognitive functions. The mini mental test is categorized under 5 main headings. It consists of 11 items including orientation (10 points), recording memory (3 points), attention and calculation (5 points), recall (3 points) and language (9 points). It is evaluated over 30 points in total. A score between 24-30 points is defined as normal, 18-23 points as mild dementia, and 17 points and below as severe dementia. The average administration time of the test is 10 minutes. Patients scoring 18 and above will be included in the study.
Expanded Disability Status Scale (EDSS) | Baseline
  The EDSS score varies between 0 and 10, and as the score increases, neurologic impairment and disability status increase in patients. While 0 is the result of neurologic evaluation obtained in a normal examination, 10 is considered as death due to MS. However, while the EDSS functions as an ambulation index in moderate and severe disability, it has been found to be highly inadequate in assessing cognitive or upper extremity functions.
Interview Form | Baseline
  All evaluations will be performed by face-to-face interview method. Individual characteristics of the patients (gender, age, height, body weight, marital status, education level, dominant extremity, smoking and alcohol consumption habits, use and type of assistive device, how many years they have been using the assistive device) and disease-related information (diagnosis year-duration, MS type, EDSS score, frequency of attacks, date of the most recent attack, medical history, family history, medications used, previous surgeries) will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: İlke KESER, Prof. Dr., Study Director — Gazi University
Locations (3):
- Turkey (Türkiye) (3):
  - Nigde Omer Halisdemir University, Niğde, Niğde Province
  - Hacettepe University, Ankara
  - Gazi University, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young CA, Mills RJ, Woolmore J, Hawkins CP, Tennant A. The unidimensional self-efficacy scale for MS (USE-MS): developing a patient based and patient reported outcome. Mult Scler. 2012 Sep;18(9):1326-33. doi: 10.1177/1352458512436592. Epub 2012 Apr 5. PMID 22492132
- [Background] Seebacher B, Mills RJ, Reindl M, Zamarian L, Kircher S, Brenneis C, Ehling R, Deisenhammer F. German translation, cultural adaptation and validation of the unidimensional self-efficacy scale for multiple sclerosis. BMC Neurol. 2021 Apr 17;21(1):163. doi: 10.1186/s12883-021-02183-y. PMID 33865337
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Background] Mills RJ, Pallant JF, Koufali M, Sharma A, Day S, Tennant A, Young CA. Validation of the Neurological Fatigue Index for stroke (NFI-Stroke). Health Qual Life Outcomes. 2012 May 15;10:51. doi: 10.1186/1477-7525-10-51. PMID 22587411